CLINICAL TRIAL: NCT06169722
Title: TDI01 for Treatment of Moderate or Severe Chronic Graft-Versus-Host Disease After Failure of at Least 1 and Not More Than 5 Lines of Systemic Therapy: an Open Label, Multi-center, ph1/2 Study
Brief Title: TDI01 Suspension in the Treatment of Chronic Graft-versus-host Disease (cGVHD))
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TDI01-YZ-101
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: GVHD, Chronic
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 200mg (Active Comparator): 200mg oral once a day
  Interventions: Drug: TDI01 suspension
- 400mg (Active Comparator): 400mg oral once a day
  Interventions: Drug: TDI01 suspension
- 200mg or 400mg (Active Comparator): 200mg or 400mg oral once a day
  Interventions: Drug: TDI01 suspension

INTERVENTIONS:
Drug: TDI01 suspension — 200mg or 400mg oral once a day

SUMMARY:
1. Phase Ib study stage:

   Primary objective: To evaluate the efficacy and safety Secondary objectives: To evaluate the population pharmacokinetic characteristics
2. Phase II study stage:

Primary objective: To evaluate the efficacy Secondary objectives: To evaluate the safety

DETAILED DESCRIPTION:
1. Phase Ib study stage:

   Primary objective: To evaluate the efficacy and safety of TDI01 suspension in treating patients with moderate or severe Chronic Graft-Versus-Host Disease after failure of at least 1 and not more than 5 lines of systemic therapy Secondary objectives: To evaluate the population pharmacokinetic characteristics of TDI01 suspension in treating patients with moderate or severe Chronic Graft-Versus-Host Disease after failure of at least 1 and not more than 5 lines of systemic therapy.
2. Phase II study stage:

Primary objective: To evaluate the efficacy of TDI01 suspension in treating patients with moderate or severe Chronic Graft-Versus-Host Disease after failure of at least 1 and not more than 5 lines of systemic therapy Secondary objectives: To evaluate the safety of TDI01 suspension in treating patients withmoderate or severe Chronic Graft-Versus-Host Disease after failure of at least 1 and not more than 5 lines of systemic therapy as well as the population pharmacokinetic characteristics of TDI01 suspension in treating these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study, sign the informed consent form, and have good compliance;
2. Subjects are aged between 18 and 75 years old, regardless of gender;
3. Within 7 days prior to the first dose, the Eastern Cooperative Oncology Group (ECOG) performance status score is 0-2;
4. Subjects are expected to survive for more than 6 months;
5. Subjects have previously received allogeneic hematopoietic stem cell transplantation;
6. Subjects have received systemic treatment for cGVHD of ≤5 lines but ≥1 line before;
7. Diagnosed with moderate to severe cGVHD based on NIH criteria, defined as follows:

   Moderate cGVHD: involvement of ≥3 organs with organ scores of 1 point, or involvement of ≥1 organ (excluding the lung) with organ scores of 2 points, or involvement of the lung with organ scores of 1 point; Severe cGVHD: involvement of ≥1 organ (excluding the lung) with organ scores of 3 points, or involvement of the lung with organ scores of 2 points or higher.
8. Diagnosed with glucocorticoid-resistant/dependent cGVHD based on NIH criteria, meeting any of the following conditions:

Subjects who have received at least 2 lines but no more than 5 lines in the past are required to have stable systemic therapy (such as corticosteroids, calcineurin inhibitors, sirolimus, mycophenolate mofetil (MMF), methotrexate, and extracorporeal phototherapy (ECP)) for at least two weeks prior to screening.

Subjects who have only received first-line glucocorticoid combined or not combined with calcineurin inhibitors in the past,Diagnosed as glucocorticoid resistant/dependent cGVHD according to NIH criteria, meeting any of the following conditions:

Subjects receiving ≥1 mg/kg prednisone (or equivalent dose of glucocorticoids) for at least 1 week but still have disease progression (glucocorticoid-resistant cGVHD); Subjects receiving ≥0.5 mg/kg/day or ≥1 mg/kg every other day prednisone (or equivalent dose of glucocorticoids) for at least 4 weeks but still have persistent disease symptoms without improvement ( glucocorticoid-resistant cGVHD); Subjects who have failed to reduce the glucocorticoid dose twice and have increased the prednisone (or equivalent dose of glucocorticoids) to >0.25 mg/kg/day (glucocorticoid-dependent cGVHD).

Exclusion Criteria:

1. The presence of recurrence of the primary disease, or having received treatment for recurrence of the primary disease after allo-HSCT（Hematopoietic stem cell transplant）, or the possible need for rapid immunosuppressive drug withdrawal as emergency treatment for early recurrence of malignant tumors; or the presence of post-transplant lymphoproliferative disorders.
2. Patients with acute GVHD and those with overlapping chronic GVHD.
3. Patients who have suffered from other malignant tumors except for the transplanted tumor within the past 3 years, with the exception of locally curable cancers (i.e., those that have already been cured), such as basal cell carcinoma or squamous cell carcinoma of the skin, cervical or breast carcinoma in situ, or superficial bladder cancer.
4. Unable to swallow medication normally, or with gastrointestinal dysfunction, or deemed by the investigator to potentially affect drug absorption.
5. The presence of active infection, including bacterial, fungal, viral (such as CMV(cytomegalovirus), EBV(epstein-barr virus), etc.) or parasitic infections that require treatment.
6. Poor diabetes control (fasting blood glucose (FBG) > 10 mmol/L).
7. Inadequate blood pressure control (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100 mmHg).
8. History of myocardial infarction within 6 months prior to planned initiation of TDI01 treatment, or arrhythmia (CTC AE(adverse event) grade 2 or higher, including QTcF ≥450ms (men), QTcF ≥470ms (women)) and congestive heart failure grade ≥2 (New York Heart Association (NYHA) classification).
9. At the time of screening, forced expiratory volume in 1 second (FEV1) ≤ 39% or NIH pulmonary symptom score of 3.
10. Received systemic treatment for cGVHD within 14 days prior to enrollment; if the dose/regimen of systemic treatment has been stable for at least 2 weeks prior to screening (corticosteroids, calcineurin inhibitors, sirolimus, mycophenolate mofetil (MMF), methotrexate, and extracorporeal photopheresis (ECP)), it is allowed.
11. Patients receiving treatment with Ibrutinib or Ruxolitinib within the past 28 days prior to the first administration of the study drug (except those who have completed washout prior to the first administration of the study drug) are excluded from participation in the study.
12. Patients who participated in other drug or device clinical trials within 4 weeks prior to the screening visit (or 5 half-lives, whichever is longer).
13. Patients receiving treatment with Warfarin or any other coumarin derivative anticoagulant, or patients with a bleeding tendency or coagulation disorder.
14. Patients with positive HBsAg and/or HBcAb and positive HBV-DNA (HBV-DNA negative patients are eligible); patients with positive HCV (hepatitis C virus) antibody and HCV-RNA copy number above the lower limit of detection. Note: Eligible patients with positive hepatitis B surface antigen or hepatitis B core antibody, and patients with hepatitis C, require continuous antiviral therapy to prevent virus activation.
15. Patients with positive HIV antibody.
16. Patients who have previously received treatment with a ROCK2 inhibitor.
17. Patients with a known history of severe allergic reactions to the study drug or its major ingredients.
18. Pregnant or breastfeeding women.
19. Patients with known alcohol or drug dependence.
20. Any other reason that the investigator believes may prevent a patient from participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Phase Ib study stage:The best overall response rate (BORR) | 24 weeks.
  The best overall response rate (BORR) at 24 weeks.
Phase Ib study stage:adverse events | 24 weeks.
  The incidence of adverse events, including treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and treatment-related adverse events (TRAEs).
Phase II study stage:The best overall response rate (BORR) | 24 weeks.
  The best overall response rate (BORR) at 24 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China